CLINICAL TRIAL: NCT03878303
Title: A Phase 1b Double-Blind, Randomized, Placebo-Controlled Study of the Safety, Pharmacokinetics and Pharmacodynamics of AC0058TA in Patients With Systemic Lupus Erythematosus (SLE)
Brief Title: Study of AC0058TA in Patients With Systemic Lupus Erythematosus (SLE)
Status: Unknown | Phase: Phase 1 | Type: Interventional
Last Known Status: Recruiting
Sponsor: ACEA Therapeutics, Inc. (Industry)
Collaborators: Hangzhou ACEA Pharmaceutical Research Co., Ltd. (Industry)
Responsible Party: Sponsor
Allocation: Randomized | Model: Parallel | Masking: Double | Purpose: Treatment
Other Study IDs: AC00582017-101
Record Dates: First submitted 2019-03-05; First posted 2019-03-18 (Actual); Last update posted 2019-03-18 (Actual); Status verified 2019-03

CONDITIONS: Systemic Lupus Erythematosus
Keywords: SLE
MeSH Terms: conditions — Lupus Erythematosus, Systemic

STUDY DESIGN:
Who Masked: Participant, Investigator
Oversight: Data Monitoring Committee: Yes | FDA-regulated Drug: Yes | FDA-regulated Device: No

ARMS (2):
- AC0058TA (Experimental): AC0058TA will be administered in 25 mg capsules orally at the following doses: 50 mg QD, 100 mg QD, 200 mg QD and 100 mg BID
  Interventions: Drug: AC0058TA
- Placebo AC0058TA (Placebo Comparator): Placebo AC0058TA will be administered orally at the equivalent dose of investigational product
  Interventions: Drug: Placebo AC0058TA

INTERVENTIONS:
Drug: AC0058TA — 25 mg capsules
  Other Names: AC0058
  Arms: AC0058TA
Drug: Placebo AC0058TA — equivalent dose of investigational product
  Other Names: Placebo
  Arms: Placebo AC0058TA

SUMMARY:
This is a Phase 1b, double blind, randomized, placebo-controlled study of the safety and tolerability, pharmacokinetics and pharmacodynamics of AC0058TA in patients with systemic lupus erythematosus (SLE).

DETAILED DESCRIPTION:
The study will be performed in adult patients with autoantibody (ANA) positive SLE, as defined by the American College of Rheumatology (ACR) 1997 criteria or System Lupus International Collaborating Clinic (SLICC) 2009 criteria who are receiving standard of care therapy for SLE.

ELIGIBILITY:
Inclusion Criteria:

1. Clinical diagnosis of SLE according to ACR 1997 criteria or 2009 SLE-SLICC criteria with ANA positive (≥ 1:40) patients who could receive hydroxychloroquine and/or steroids treatment.
2. Adequate hematopoietic function, including:

   * Platelet count > 75 × 10^9/L
   * Leukocyte ≥ 2.0 × 10^9/L including CD19+ B cell counts of at least 50/μL
   * Hemoglobin ≥ 10 g/dL
3. Adequate liver function

   * Bilirubin: < 1.2 X upper limit of normal (ULN)
   * AST: < 1.2 X upper limit of normal (ULN)
   * ALT: < 1.2 X upper limit of normal (ULN)
4. Adequate renal function:

   a. BUN and creatinine:< 1.5 X upper limit of normal (ULN)
5. Female of reproductive potential must agree to use two forms of contraception during screening, during the study, and for at least 30 days after the last dose of AC0058TA.
6. Able to provide written informed consent in accordance with federal, local, and institutional guidelines.

Exclusion Criteria:

1. Active central nervous system (CNS) lupus (including seizures, psychosis, organic brain syndrome, cerebrovascular accident [CVA], cerebritis or CNS vasculitis) or active bleeding disorder within 60 days prior to the first day of study treatment.
2. Clinical evidence of significant unstable or uncontrolled acute or chronic diseases other than SLE which, in the opinion of the investigator, could confound the results of the study, put the patient at undue risk, or interferes with protocol adherence, or a subject's ability to give informed consent.
3. History or presence of congestive heart failure (New York Heart Association [NYHA]Class III to IV), symptomatic ischemia, clinically significant conduction abnormalities uncontrolled by conventional intervention, or myocardial infarction within 6 months prior to the first day of study treatment.
4. Have severe lupus complications (Acute Lupus Pneumonitis, Diffuse Alveolar Hemorrhage, Chronic Interstitial Pneumonia, Pulmonary Hypertension, Pulmonary Embolism) severe lupus gastrointestinal diseases (Lupus Mesenteric Vasculitis, Protein-Losing Enteropathy, Pancreatitis, Intestinal Pseudo-Obstruction).
5. History of any bleeding disorder secondary to SLE.
6. Have active, severe lupus kidney disease WHO III-V (Rapidly Progressive Glomerulonephritis, Nephrotic Syndrome, Renal Tubular Acidosis, Renal Insufficiency), proteinuria > 500 mg/day.
7. Acute or chronic infections requiring systemic antibiotic, antifungal, or antiviral therapy within 60 days of the first day of study treatment.
8. Known HIV infection or positive for hepatitis B virus infection (HBsAg positive, HBeAg, HBeAb or HBcAb positive and HBV DNA positive) or hepatitis C antibody positive (HCV RNA positive).
9. Primary immunodeficiency other than complement deficiencies.
10. Active or latent tuberculosis within 6 months prior to the first day of study treatment.
11. Receipt of a live-attenuated vaccine within 2 months prior to screening.
12. Within 2 weeks prior to screening：Use of injectable corticosteroids.
13. Within 2 months prior to screening: use of abatacept, anti-tumor necrosis factor alpha agents, intravenous immunoglobulin, plasmapheresis, mycophenolate, MTX and leflunomide or therapies not otherwise specified in protocol.
14. Use of cyclophosphamide or chlorambucil within five half-lives of screening.
15. Use of rituximab, belimumab, or any other B cell-depleting or modulating therapies within 6 months of screening.
16. Female patients who are pregnant or breastfeeding.
17. Use of an investigational therapeutics within 30 days or 5 half-lives prior to screening, whichever is greater.
18. Has a positive pregnancy test result at Screening or Check-in (females only).
19. Women with childbearing potential are defined as all women who are physiologically able to have a pregnancy, unless they are using an efficient contraceptive method during treatment and within 30 days after discontinuation of treatment as below.

    1. Complete abstinence (if this is in line with the subject's preferred and usual lifestyle). Periodic abstinence (e.g., calendaring method, ovulation method, symptomatic body temperature method, post-ovulation method) and in vitro ejaculation are unacceptable contraceptive methods.
    2. Patients who have received female sterilization (bilateral ovariectomy with or without hysterectomy) or tubal ligation for at least 6 weeks prior to study treatment. In case of only unilateral ovariectomy, female fertility status must be confirmed by follow-up assessment of hormone levels.
    3. Combination of the following two methods:

       * Intrauterine device (IUD) or intrauterine system (IUS).
       * Barrier contraceptive methods: condoms or cervical cap (diaphragm or cervical cap) coated with spermicidal foam/gel/cream/vaginal suppositories. If women use oral contraceptives only, they should use the same contraceptives at a stable dose for at least 3 months before starting the study treatment.
    4. If women have at least 12 months of natural amenorrhea and are clinically compatible (e.g., at the corresponding age, with a history of vasomotor symptoms or received bilateral ovariectomy with or without hysterectomy, they are regarded as postmenopausal women with no childbearing potential. In case of only unilateral ovariectomy, female fertility status must be confirmed by follow-up assessment of hormone levels before the women can be considered to have no childbearing potential.
20. Men who have sexual intercourse unless they use a condom during sexual intercourse and must not donate sperm from the first dose of study drug until 30 days after discontinuation of treatment and do not impregnate their sexual partners during the period. Vasectomized males are also required to use condoms to prevent the transmission of drugs through semen.
21. Subject who, in the opinion of the Investigator, should not participate in this study.

Ages: 18 Years to 75 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Enrollment: 32 (Estimated)
Dates: Start 2018-11-28 (Actual); Primary Completion 2020-12 (Estimated); Study Completion 2021-12 (Estimated)

PRIMARY OUTCOMES:
Incidence of Treatment-Emergent Adverse Events and Serious Adverse Events | Measured up to 12 weeks

SECONDARY OUTCOMES:
Maximum Plasma Concentration and Area Under the Curve | Measured on Day 1, Day 28, and Day 84
Pharmacodynamics of AC0058TA: Bruton's tyrosine kinase (BTK) occupancy (% occupancy) | Measured on Day 1, Day 28, and Day 84
Pharmacodynamics of AC0058TA: serum antidsDNA antibodies, ANAs, complement (C3 and C4) and B-cell markers | Measured on Day 1, Day 28, and Day 84

CONTACTS AND LOCATIONS:
Overall Officials: Roy Fleischmann, MD MACR, Principal Investigator — Metroplex Clinical Research Center
Locations (1):
- Metroplex Clinical Research Center, Dallas, Texas, United States